CLINICAL TRIAL: NCT06181500
Title: Home-Based Exercise in Primary Progressive Aphasia: A Pilot Study
Brief Title: Home-Based Exercise in Primary Progressive Aphasia (HEPPA)
Acronym: HEPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Louis Bherer, Director of the EPIC Center and Scientist, Montreal Heart Institute, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-33-2022-3114
Record Dates: First submitted 2023-11-19; First posted 2023-12-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-12

CONDITIONS: Primary Progressive Aphasia; Neurodegenerative Diseases; Logopenic Progressive Aphasia; Semantic Dementia; Non-fluent Aphasia
Keywords: Primary Progressive Aphasia; Home-Based Exercise Intervention; Pilot Study
MeSH Terms: conditions — Aphasia, Primary Progressive; Neurodegenerative Diseases; Frontotemporal Dementia; Aphasia, Broca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home-based multicomponent exercise intervention program (Experimental)
  Interventions: Other: Home-based multicomponent exercise intervention program

INTERVENTIONS:
Other: Home-based multicomponent exercise intervention program — A novel home-based multicomponent exercise intervention program was designed using a multimodal training circuit. This 24-week circuit program was created to improve functional (resistance) and aerobic health. Participants will be asked to train two to three times a week for 45 minutes. They will be supervised via videoconference by a trained kinesiologist from the EPIC Center at the Montreal Heart Institute. If desired, participants can complete their exercises with a partner, friend, or relative to facilitate communication. Participants will be asked to document the perceived intensity of their exercises in a booklet after each workout. The perceived intensity of their exercises will be measured by a validated effort perception scale graduated from 0 to 10 (Borg scale; Williams, 2017). Progressions will increase every five weeks and will be subject to modification if not properly tolerated or if found to be below a 3 on the Borg rate of perceived exertion scale (moderate intensity).

SUMMARY:
This pilot study aims to evaluate the feasibility of a novel home-based multicomponent exercise program in adults clinically diagnosed with Primary Progressive Aphasia

DETAILED DESCRIPTION:
Exercise is known to induce changes in brain neuroplasticity in the elderly and is thought to have a protective effect against cognitive decline in patients already suffering from neurodegenerative diseases. While the benefits of exercise in the context of mild cognitive impairment and Alzheimer's disease have been extensively studied, little information is available on the potential benefits of exercise for other atypical neurodegenerative diseases, such as primary progressive aphasia (PPA). A multimodal exercise intervention (combination of aerobic and resistance exercises) could potentially slow overall cognitive decline in PPA, which is characterized by a gradual and isolated dissolution of language function, by promoting neurogenesis and neuroplasticity. In healthy but inactive older adults, exercise increases grey and white matter volume in prefrontal and temporal cortical regions, which are specifically impaired in PPA and play an important role in executive functions, episodic memory and language skills. Exercise could thus modulate certain executive, memory and language difficulties generally observed in this clinical population. This pilot study aims to evaluate the feasibility of a novel home-based multicomponent exercise program in adults clinically diagnosed with any of the three main variants of PPA (semantic, non-fluent/agrammatic or logopenic). The feasibility outcomes will be based on: 1) total recruitment and recruitment rate, 2) program completion rate, 3) compliance and 4) participants' ability to train at home with or without a caregivers' presence. A minimum of 12 participants will be recruited through McGill University's Douglas Research Institute and will complete a 6-month home-based multimodal intervention program. They will train two to three times a week for 45 minutes and be supervised via videoconference by a kinesiologist from the EPIC Center at the Montreal Heart Institute. If desired, participants will be accompanied by a partner, close friend, or relative to facilitate communication, especially if they have difficulty understanding instructions or expressing themselves. To assess changes in cognition, physical and psychological functions, participants will complete neuropsychological and functional assessments in-person at baseline. These assessments will also be completed at three and six months post-intervention. The knowledge gained from this pilot project will be used to assess the feasibility of a full randomized control trial aimed at assessing the effects of multimodal exercise intervention in PPA patients. Ultimately, an increased understanding of the potential beneficial effects of physical exercise in PPA will allow for more tailored rehabilitative approaches in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Primary Progressive Aphasia
* Fluent in French or English
* Able to read, understand and sign the information and consent form
* Have access to the internet
* Have access to a tablet (i.e. iPad or Android) or a computer

Exclusion Criteria:

* Any absolute and relative contraindication to exercise testing and/or physical training (e.g., any severe musculoskeletal disease impairing their mobility)
* Any severe respiratory disease (e.g., asthma, COPD, COVID-19)
* Any severe exercise intolerance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the total recruitment rate of a 6-month exercise intervention in individuals with Primary Progressive Aphasia | 6 months post-intervention
  Total recruitment (number of participants screened compared to final enrollments)
Evaluate the recruitment rate of a 6-month exercise intervention in individuals with Primary Progressive Aphasia | 6 months post-intervention
  Recruitment rate (number of participants that can be enrolled per month)
Evaluate the program completion rate of a 6-month exercise intervention in individuals with Primary Progressive Aphasia | 6 months post-intervention
  Program completion rate (number of participants that completed their in-person evaluations as well as the home-based interventions after 6 months compared to the participants enrolled)
Evaluate the compliance rate of a 6-month exercise intervention in individuals with Primary Progressive Aphasia | 6 months post-intervention
  Compliance (total number of in-person evaluations and home-based training sessions attended compared to the maximum possible)
Evaluate the satisfaction of a 6-month exercise intervention in individuals with Primary Progressive Aphasia | 6 months post-intervention
  Satisfaction (feedback given by the participants and their caregivers will be considered using a satisfaction questionnaire and qualitative feedback). Ability to train at home with or without their caregivers' presence will also be taken into account.

SECONDARY OUTCOMES:
Document changes in general cognitive functioning | Baseline and 6 months post-intervention
  Participants will complete the Montreal Cognitive Assessment (scores range from 0-28, with a higher score indicating better cognitive functioning).
Document changes in auditory long-term memory | Baseline and 6 months post-intervention
  Participants will complete the Rey auditory verbal learning test (scores range from 0-15, with a higher score indicating a better auditory long-term memory).
Document changes in visual long-term memory | Baseline and 6 months post-intervention
  Participants will complete the Rey-Osterrieth complex figure test (scores range from 0-36, with a higher score indicating a better visual long-term memory).
Document changes in verbal working memory | Baseline and 6 months post-intervention
  Participants will complete the forward and backward digit span subtasks of the Wechsler Adult Intelligence Scale-IV (scores range from 0-32, with a higher number indicating a better score).
Document changes in visual working memory | Baseline and 6 months post-intervention
  Participants will complete the spatial span subtask of the Wechsler Memory Scale-III (scores range from 0-32, with a higher number indicating a better score).
Document changes in nonverbal fluency | Baseline and 6 months post-intervention
  Participants will complete the Ruff figure fluency test (scores are based on the total number of figures drawn, with a higher number indicating a better score).
Document changes in verbal fluency | Baseline and 6 months post-intervention
  Participants will complete phonemic and semantic fluency tasks (scores are based on the total number of words given, with a higher number indicating a better score).
Document changes in reading comprehension | Baseline and 6 months post-intervention
  Participants will complete the Chapman-Cook (scores range from 0-30, with a higher score indicating better reading comprehension).
Document changes in writing ability | Baseline and 6 months post-intervention
  Participants will complete the Bernard Croisile dictation task (scores range from 0-18, with a higher score indicating better writing ability).
Document changes in auditory comprehension | Baseline and 6 months post-intervention
  Participants will complete the Boston Diagnostic Aphasia Examination (BDAE) subtasks: word, body part, commands, story comprehension, and the word-picture matching (scores range from 0-36, with higher scores indicating better auditory comprehension).
Document changes in oral expression | Baseline and 6 months post-intervention
  Participants will complete the word/sentence repetition subtasks from the Boston Diagnostic Aphasia Examination (BDAE) (scores range from 0-14, with higher scores indicating better oral expression).
Document changes in lexical retrieval | Baseline and 6 months post-intervention
  Participants will complete the Boston Naming Test (scores range from 0-30, with a higher score indicating better lexical retrieval).
Document changes in executive functions and processing speed | Baseline and 6 months post-intervention
  Participants will complete validated neuropsychological tests and iPad tests (scores are measured in milliseconds, with lower reaction times indicating faster processing speeds).
Document changes in endurance | Baseline and 6 months post-intervention
  Endurance will be assessed with a 6 min walking test (scores are measured in the number of meters walked, with a higher number of meters indicating a better score).
Document change in balance performance | Baseline and 6 months post-intervention
  Balance performance will be assessed with a timed one-leg standing test (scores are measured in seconds, with a higher time indicating a better score).
Document change in upper limb muscle strength | Baseline and 6 months post-intervention
  Upper limb muscle strength will be assessed with a grip strength test (scores are measured with the maximum force/tension generated by one's forearm muscles, with a higher kilogram indicating a better score).
Document change in lower limb muscle strength | Baseline and 6 months post-intervention
  Lower limb muscle strength will be assessed with a timed Sit-to-Stand test (scores are measured in seconds, with a lower time indicating a better score).
Document changes in walking speed | Baseline and 6 months post-intervention
  Walking speed will be assessed with a 10-meter walking test (scores are measured in seconds, with a lower time indicating a better score).
Document changes functional mobility | Baseline and 6 months post-intervention
  Functional mobility will be assessed with the Timed up and Go test (scores are measured in seconds, with a lower time indicating a better score).
Document changes in cardiorespiratory fitness | Baseline and 6 months post-intervention
  Cardiorespiratory fitness will be assessed with the Matthews cardiorespiratory fitness questionnaire (the score is an estimation of individual VO2 max (ml.kg.min) and ranges from 15-50, with a higher score indicating a higher VO2max).

OTHER OUTCOMES:
Document changes in quality-of-life | Baseline and 6 months post-intervention
  12-Item Short Form Health Survey. This questionnaire gives two scores - a mental component scale (MCS) and a physical component scale (PCS) score. Results are reported as Z-scores (mean of 50 and standard deviation of 10) and so each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Document changes in depressive symptomatology | Baseline and 6 months post-intervention
  Geriatric Depression Scale questionnaire (scores range from 0-30, with a higher score indicating larger depressive symptomatology).
Document changes in anxiety | Baseline and 6 months post-intervention
  State-Trait Anxiety Inventory questionnaire (scores range from 20-80, with a higher score indicating higher anxiety).
Document changes in perceived stress | Baseline and 6 months post-intervention
  Perceived Stress Scale questionnaire (scores range from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe).
Document changes in sleep quality | Baseline and 6 months post-intervention
  Pittsburg Sleep Quality Index questionnaire (scores range from 0-21, with a higher score indicating worse sleep quality).
Document changes in risk of sleep apnea | Baseline and 6 months post-intervention
  Using the Berlin Questionnaire, participants are classified into high risk or low risk based on their responses to the individual items and their overall scores in the symptom categories (high risk = if there are 2 or more categories where the score is positive/ low risk = if there are only 1 or no categories where the score is positive).
Document changes in self-reported physical activity | Baseline and 6 months post-intervention
  Physical Activity Scale for the Elderly questionnaire (scores range from 0-400, with a higher score indicating better level of physical activity).
Document changes in neuropsychiatric symptoms | Baseline and 6 months post-intervention
  The Neuropsychiatric Inventory-Questionnaire is completed by the participants' caregiver (scores range from 0-36 for symptom severity and from 0-60 for the caregiver's distress, with higher scores indicating higher severity/distress).
Document Cognitive Reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (scores range from 0-26, with a higher score indicating a greater cognitive reserve).
Document perceived social support | Baseline
  Lubben Social Network Scale questionnaire (scores range from 0-30, with a higher score indicating more social engagement)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, Principal Investigator — Centre ÉPIC, Institut de cardiologie de Montréal
Locations (2):
- Canada (2):
  - Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec
  - McGill University Research Centre for Studies in Aging (MCSA), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angevaren M, Vanhees L, Wendel-Vos W, Verhaar HJ, Aufdemkampe G, Aleman A, Verschuren WM. Intensity, but not duration, of physical activities is related to cognitive function. Eur J Cardiovasc Prev Rehabil. 2007 Dec;14(6):825-30. doi: 10.1097/HJR.0b013e3282ef995b. PMID 18043306
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Plymate SR, Fishel MA, Watson GS, Cholerton BA, Duncan GE, Mehta PD, Craft S. Effects of aerobic exercise on mild cognitive impairment: a controlled trial. Arch Neurol. 2010 Jan;67(1):71-9. doi: 10.1001/archneurol.2009.307. PMID 20065132
- [Background] Bherer L, Erickson KI, Liu-Ambrose T. A review of the effects of physical activity and exercise on cognitive and brain functions in older adults. J Aging Res. 2013;2013:657508. doi: 10.1155/2013/657508. Epub 2013 Sep 11. PMID 24102028
- [Background] Blondell SJ, Hammersley-Mather R, Veerman JL. Does physical activity prevent cognitive decline and dementia?: A systematic review and meta-analysis of longitudinal studies. BMC Public Health. 2014 May 27;14:510. doi: 10.1186/1471-2458-14-510. PMID 24885250
- [Background] Borst SE, De Hoyos DV, Garzarella L, Vincent K, Pollock BH, Lowenthal DT, Pollock ML. Effects of resistance training on insulin-like growth factor-I and IGF binding proteins. Med Sci Sports Exerc. 2001 Apr;33(4):648-53. doi: 10.1097/00005768-200104000-00021. PMID 11283443
- [Background] Casaletto KB, Staffaroni AM, Wolf A, Appleby B, Brushaber D, Coppola G, Dickerson B, Domoto-Reilly K, Elahi FM, Fields J, Fong JC, Forsberg L, Ghoshal N, Graff-Radford N, Grossman M, Heuer HW, Hsiung GY, Huey ED, Irwin D, Kantarci K, Kaufer D, Kerwin D, Knopman D, Kornak J, Kramer JH, Litvan I, Mackenzie IR, Mendez M, Miller B, Rademakers R, Ramos EM, Rascovsky K, Roberson ED, Syrjanen JA, Tartaglia MC, Weintraub S, Boeve B, Boxer AL, Rosen H, Yaffe K; ARTFL/LEFFTDS Study. Active lifestyles moderate clinical outcomes in autosomal dominant frontotemporal degeneration. Alzheimers Dement. 2020 Jan;16(1):91-105. doi: 10.1002/alz.12001. PMID 31914227
- [Background] Cassilhas RC, Viana VA, Grassmann V, Santos RT, Santos RF, Tufik S, Mello MT. The impact of resistance exercise on the cognitive function of the elderly. Med Sci Sports Exerc. 2007 Aug;39(8):1401-7. doi: 10.1249/mss.0b013e318060111f. PMID 17762374
- [Background] Cheng ST, Chow PK, Song YQ, Yu EC, Chan AC, Lee TM, Lam JH. Mental and physical activities delay cognitive decline in older persons with dementia. Am J Geriatr Psychiatry. 2014 Jan;22(1):63-74. doi: 10.1016/j.jagp.2013.01.060. Epub 2013 Feb 6. PMID 23582750
- [Background] Colcombe SJ, Erickson KI, Scalf PE, Kim JS, Prakash R, McAuley E, Elavsky S, Marquez DX, Hu L, Kramer AF. Aerobic exercise training increases brain volume in aging humans. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1166-70. doi: 10.1093/gerona/61.11.1166. PMID 17167157
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Duffy JR, Strand EA, Clark H, Machulda M, Whitwell JL, Josephs KA. Primary progressive apraxia of speech: clinical features and acoustic and neurologic correlates. Am J Speech Lang Pathol. 2015 May;24(2):88-100. doi: 10.1044/2015_AJSLP-14-0174. PMID 25654422
- [Background] Eikelboom WS, Janssen N, Jiskoot LC, van den Berg E, Roelofs A, Kessels RPC. Episodic and working memory function in Primary Progressive Aphasia: A meta-analysis. Neurosci Biobehav Rev. 2018 Sep;92:243-254. doi: 10.1016/j.neubiorev.2018.06.015. Epub 2018 Jun 18. PMID 29928907
- [Background] Foxe D, Irish M, Hu A, Carrick J, Hodges JR, Ahmed RM, Burrell JR, Piguet O. Longitudinal cognitive and functional changes in primary progressive aphasia. J Neurol. 2021 May;268(5):1951-1961. doi: 10.1007/s00415-020-10382-9. Epub 2021 Jan 8. PMID 33417000
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Gorno-Tempini ML, Dronkers NF, Rankin KP, Ogar JM, Phengrasamy L, Rosen HJ, Johnson JK, Weiner MW, Miller BL. Cognition and anatomy in three variants of primary progressive aphasia. Ann Neurol. 2004 Mar;55(3):335-46. doi: 10.1002/ana.10825. PMID 14991811
- [Background] Haeger A, Costa AS, Schulz JB, Reetz K. Cerebral changes improved by physical activity during cognitive decline: A systematic review on MRI studies. Neuroimage Clin. 2019;23:101933. doi: 10.1016/j.nicl.2019.101933. Epub 2019 Jul 16. PMID 31491837
- [Background] Harris JM, Saxon JA, Jones M, Snowden JS, Thompson JC. Neuropsychological differentiation of progressive aphasic disorders. J Neuropsychol. 2019 Jun;13(2):214-239. doi: 10.1111/jnp.12149. Epub 2018 Feb 8. PMID 29424041
- [Background] Heyn P, Abreu BC, Ottenbacher KJ. The effects of exercise training on elderly persons with cognitive impairment and dementia: a meta-analysis. Arch Phys Med Rehabil. 2004 Oct;85(10):1694-704. doi: 10.1016/j.apmr.2004.03.019. PMID 15468033
- [Background] Holthoff VA, Marschner K, Scharf M, Steding J, Meyer S, Koch R, Donix M. Effects of physical activity training in patients with Alzheimer's dementia: results of a pilot RCT study. PLoS One. 2015 Apr 17;10(4):e0121478. doi: 10.1371/journal.pone.0121478. eCollection 2015. PMID 25884637
- [Background] Kolb, B., & Whishaw, I. Q. (2009). Fundamentals of human neuropsychology. Macmillan.
- [Background] Kwak YS, Um SY, Son TG, Kim DJ. Effect of regular exercise on senile dementia patients. Int J Sports Med. 2008 Jun;29(6):471-4. doi: 10.1055/s-2007-964853. Epub 2007 Nov 30. PMID 18050054
- [Background] Langlois F, Vu TT, Chasse K, Dupuis G, Kergoat MJ, Bherer L. Benefits of physical exercise training on cognition and quality of life in frail older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):400-4. doi: 10.1093/geronb/gbs069. Epub 2012 Aug 28. PMID 22929394
- [Background] Mandelli ML, Vitali P, Santos M, Henry M, Gola K, Rosenberg L, Dronkers N, Miller B, Seeley WW, Gorno-Tempini ML. Two insular regions are differentially involved in behavioral variant FTD and nonfluent/agrammatic variant PPA. Cortex. 2016 Jan;74:149-57. doi: 10.1016/j.cortex.2015.10.012. Epub 2015 Nov 14. PMID 26673947
- [Background] Marques-Aleixo I, Beleza J, Sampaio A, Stevanovic J, Coxito P, Goncalves I, Ascensao A, Magalhaes J. Preventive and Therapeutic Potential of Physical Exercise in Neurodegenerative Diseases. Antioxid Redox Signal. 2021 Mar 10;34(8):674-693. doi: 10.1089/ars.2020.8075. Epub 2020 Apr 24. PMID 32159378
- [Background] Marshall CR, Hardy CJD, Volkmer A, Russell LL, Bond RL, Fletcher PD, Clark CN, Mummery CJ, Schott JM, Rossor MN, Fox NC, Crutch SJ, Rohrer JD, Warren JD. Primary progressive aphasia: a clinical approach. J Neurol. 2018 Jun;265(6):1474-1490. doi: 10.1007/s00415-018-8762-6. Epub 2018 Feb 1. PMID 29392464
- [Background] Matthews CE, Heil DP, Freedson PS, Pastides H. Classification of cardiorespiratory fitness without exercise testing. Med Sci Sports Exerc. 1999 Mar;31(3):486-93. doi: 10.1097/00005768-199903000-00019. PMID 10188755
- [Background] Mesulam MM. Primary progressive aphasia. Ann Neurol. 2001 Apr;49(4):425-32. PMID 11310619
- [Background] Meyer AM, Snider SF, Campbell RE, Friedman RB. Phonological short-term memory in logopenic variant primary progressive aphasia and mild Alzheimer's disease. Cortex. 2015 Oct;71:183-9. doi: 10.1016/j.cortex.2015.07.003. Epub 2015 Jul 16. PMID 26232551
- [Background] Migliaccio R, Agosta F, Rascovsky K, Karydas A, Bonasera S, Rabinovici GD, Miller BL, Gorno-Tempini ML. Clinical syndromes associated with posterior atrophy: early age at onset AD spectrum. Neurology. 2009 Nov 10;73(19):1571-8. doi: 10.1212/WNL.0b013e3181c0d427. PMID 19901249
- [Background] Sampaio A, Marques EA, Mota J, Carvalho J. Effects of a multicomponent exercise program in institutionalized elders with Alzheimer's disease. Dementia (London). 2019 Feb;18(2):417-431. doi: 10.1177/1471301216674558. Epub 2016 Oct 18. PMID 27756836
- [Background] Sanders LMJ, Hortobagyi T, Karssemeijer EGA, Van der Zee EA, Scherder EJA, van Heuvelen MJG. Effects of low- and high-intensity physical exercise on physical and cognitive function in older persons with dementia: a randomized controlled trial. Alzheimers Res Ther. 2020 Mar 19;12(1):28. doi: 10.1186/s13195-020-00597-3. PMID 32192537
- [Background] Sebastian R, Thompson CB, Wang NY, Wright A, Meyer A, Friedman RB, Hillis AE, Tippett DC. Patterns of Decline in Naming and Semantic Knowledge in Primary Progressive Aphasia. Aphasiology. 2018;32(9):1010-1030. doi: 10.1080/02687038.2018.1490388. Epub 2018 Jun 28. PMID 30613121
- [Background] Siddiqui SV, Chatterjee U, Kumar D, Siddiqui A, Goyal N. Neuropsychology of prefrontal cortex. Indian J Psychiatry. 2008 Jul;50(3):202-8. doi: 10.4103/0019-5545.43634. PMID 19742233
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924
- [Background] Spinelli EG, Mandelli ML, Miller ZA, Santos-Santos MA, Wilson SM, Agosta F, Grinberg LT, Huang EJ, Trojanowski JQ, Meyer M, Henry ML, Comi G, Rabinovici G, Rosen HJ, Filippi M, Miller BL, Seeley WW, Gorno-Tempini ML. Typical and atypical pathology in primary progressive aphasia variants. Ann Neurol. 2017 Mar;81(3):430-443. doi: 10.1002/ana.24885. Epub 2017 Mar 20. PMID 28133816
- [Background] Tan ZS, Spartano NL, Beiser AS, DeCarli C, Auerbach SH, Vasan RS, Seshadri S. Physical Activity, Brain Volume, and Dementia Risk: The Framingham Study. J Gerontol A Biol Sci Med Sci. 2017 Jun 1;72(6):789-795. doi: 10.1093/gerona/glw130. PMID 27422439
- [Background] Tarazona-Santabalbina FJ, Gomez-Cabrera MC, Perez-Ros P, Martinez-Arnau FM, Cabo H, Tsaparas K, Salvador-Pascual A, Rodriguez-Manas L, Vina J. A Multicomponent Exercise Intervention that Reverses Frailty and Improves Cognition, Emotion, and Social Networking in the Community-Dwelling Frail Elderly: A Randomized Clinical Trial. J Am Med Dir Assoc. 2016 May 1;17(5):426-33. doi: 10.1016/j.jamda.2016.01.019. Epub 2016 Mar 3. PMID 26947059
- [Background] Teixeira CVL, Ribeiro de Rezende TJ, Weiler M, Magalhaes TNC, Carletti-Cassani AFMK, Silva TQAC, Joaquim HPG, Talib LL, Forlenza OV, Franco MP, Nechio PE, Fernandes PT, Cendes F, Balthazar ML. Cognitive and structural cerebral changes in amnestic mild cognitive impairment due to Alzheimer's disease after multicomponent training. Alzheimers Dement (N Y). 2018 Aug 30;4:473-480. doi: 10.1016/j.trci.2018.02.003. eCollection 2018. PMID 30258976
- [Background] Teixeira CV, Rezende TJ, Weiler M, Nogueira MH, Campos BM, Pegoraro LF, Vicentini JE, Scriptore G, Cendes F, Balthazar ML. Relation between aerobic fitness and brain structures in amnestic mild cognitive impairment elderly. Age (Dordr). 2016 Jun;38(3):51. doi: 10.1007/s11357-016-9912-3. Epub 2016 Apr 23. PMID 27106271
- [Background] Venegas-Sanabria LC, Martinez-Vizcaino V, Cavero-Redondo I, Chavarro-Carvajal DA, Cano-Gutierrez CA, Alvarez-Bueno C. Effect of physical activity on cognitive domains in dementia and mild cognitive impairment: overview of systematic reviews and meta-analyses. Aging Ment Health. 2021 Nov;25(11):1977-1985. doi: 10.1080/13607863.2020.1839862. Epub 2020 Nov 4. PMID 33143444
- [Background] WHO. (2020). WHO guidelines on physical activity and sedentary behaviour: at a glance. Williams, N. (2017). The Borg rating of perceived exertion (RPE) scale. Occupational Medicine, 67(5), 404-405
- [Background] Zhu L, Li L, Wang L, Jin X, Zhang H. Physical Activity for Executive Function and Activities of Daily Living in AD Patients: A Systematic Review and Meta-Analysis. Front Psychol. 2020 Dec 3;11:560461. doi: 10.3389/fpsyg.2020.560461. eCollection 2020. PMID 33343442